CLINICAL TRIAL: NCT01513707
Title: The Effects of Pre-transplant Dialysis Modality on Post-transplant Events
Acronym: PDMP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ha Young Oh (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor-Investigator, Ha Young Oh, professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Other Study IDs: 2011-12-005
Record Dates: First submitted 2012-01-16; First posted 2012-01-20 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Delayed Function of Renal Transplant; Primary Nonfunction of Renal Transplant; Acute Rejection of Renal Transplant
Keywords: kidney transplantation; hemodialysis; peritoneal dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hemodialysis group: Hemodialysis group
- peritoneal dialysis group: peritoneal dialysis group

SUMMARY:
This is a prospective, multicenter, comparative, parallel-group, observational study. There will be 2 cohorts according to pre-transplant dialysis modality (hemodialysis or peritoneal dialysis). In each cohort, subjects will be observed for 12 months. Approximately, 1040 subjects will be enrolled from 8 transplant centers.

Subjects will be enrolled consecutively until the number of subjects in peritoneal dialysis group has been 260. It will take 2 years. In this period, the number of subject in hemodialysis group enrolled in this study will be 780. After finishing the observation of all subjects, to balance clinical and demographic baseline characteristics between the two groups, subjects will be selected in each cohort with 1:1 matched using propensity score method. And then primary and secondary endpoints will be compared between two groups.

DETAILED DESCRIPTION:
1. STUDY OBJECTIVES AND ENDPOINTS 1.1. Objectives

The primary objective of this study is:

• To compare the incidence of composite outcomes (delayed graft function, functional delayed graft function, primary nonfunction, biopsy-proven acute rejection) of pre-transplant dialysis modality hemodialysis versus peritoneal in recipients of first renal allografts at 1 year posttransplant.

The secondary objectives of this study are:

* To compare the incidence of delayed graft function and functional delayed graft function of pre-transplant dialysis modality hemodialysis versus peritoneal in recipients of first renal allografts at 1 year posttransplant;
* To compare the incidence of composite outcomes biopsy-proven acute rejection of pre-transplant dialysis modality hemodialysis versus peritoneal in recipients of first renal allografts at 1 year posttransplant;
* To compare the incidence of primary nonfunction of pre-transplant dialysis modality hemodialysis versus peritoneal in recipients of first renal allografts at 1 year posttransplant;
* To evaluate the effect of hemodialysis or peritoneal dialysis on graft function in terms of longitudinal change of eGFR calculated with abbreviated MDRD equation at Weeks 8, 16, 24, 32, 40, and 48 after renal transplant;
* To compare the incidence and the duration of hospitalization after kidney transplantation of pre-transplant dialysis modality hemodialysis versus peritoneal in recipients of first renal allografts at 1 year posttransplant;
* To compare the graft loss and subject death rate of pre-transplant dialysis modality hemodialysis versus peritoneal in recipients of first renal allografts at 1 year posttransplant.

1.2. Endpoints

Primary endpoint:

* Composite outcome including;

  1. Delayed graft function (defined as the need for dialysis in the first week after transplantation)
  2. Functional DGF (defined as the absence of a decrease in serum creatinine level by a minimum of 10% per day during 3 consecutive days in the first postoperative week, not including patients in whom acute rejection, calcineurin inhibitor toxicity, or both, developed within the first week
  3. Primary nonfunction (defined as the kidney never achieving function after transplantation)
  4. Biopsy proven acute rejection (defined as scute rejection, confirmed by allograft biopsy)

     Secondary endpoints:
* eGFR (calculated with abbreviated MDRD equation at Weeks 8, 16, 24, 32, 40 and 48 after renal transplant)
* Hospitalization after kidney transplant (any cause, duration)
* Delayed graft function, functional DGF, Primary nonfunction, biopsy proven acute rejection (definition of each endpoint is described above)
* Graft loss (return to long-term dialysis)
* Subject death (any cause)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have end-stage renal disease, have been on one renal replacement therapy (hemodialysis or peritoneal dialysis) for > 6 months ( Who had been on hemodialysis for at least 6 months before renal transplant for the hemodialysis group; Who had been on peritoneal dialysis for at least 6 months before renal transplant for the peritoneal dialysis group ), and are scheduled to receive a first kidney transplant from a deceased donor, a living-related donor, or a living-unrelated donor.
2. Between the ages of 20 and 70 years, inclusive.
3. Either female or male adults
4. Subjects must be willing and able to provide written personal information consent with evidence of a personally signed and dated personal information consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Subjects who had combined dialysis (hemodialysis + peritoneal dialysis simultaneously).
2. Subjects who are recipients for multiple organ transplant.
3. Subjects scheduled for non-heart beating donor transplantation.
4. Subjects scheduled for transplantation using desensitization (plasmapheresis + Rituximab) process.
5. Subjects with evidence of active infection.
6. Women of childbearing potential who are either pregnant, lactating, planning to become pregnant in the next 12 months. Women of childbearing potential must be willing to agree to contraceptive practices.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 1040 (Estimated)
Dates: Start 2011-12-22 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
composite outcomes (delayed graft function, functional delayed graft function, primary nonfunction, biopsy-proven acute rejection) | 1 year posttransplant
  1. Delayed graft function
  2. Functional DGF (defined as the absence of a decrease in serum creatinine level by a minimum of 10% per day during 3 consecutive days in the first postoperative week, not including patients in whom acute rejection, calcineurin inhibitor toxicity, or both, developed within the first week
  3. Primary nonfunction
  4. Biopsy proven acute rejection

SECONDARY OUTCOMES:
eGFR | 1 year
  • eGFR (calculated with abbreviated MDRD equation at Weeks 8, 16, 24, 32, 40 and 48 after renal transplant)
Hospitalization | 1 year
  • Hospitalization after kidney transplant (any cause, duration)
graft loss | 1 year
  • Graft loss (return to long-term dialysis)
Subject death | 1 year
  • Subject death (any cause)

CONTACTS AND LOCATIONS:
Overall Officials: Hayoung Oh, Principal Investigator — South Korea Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided